CLINICAL TRIAL: NCT03046615
Title: Intraoperative Non-invasive Eye Movement Monitoring
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jamie J. Van Gompel, Associate Professor of Neurosurgery and Otolaryngology, Mayo Clinic
Other Study IDs: 16-010266
Record Dates: First submitted 2017-02-01; First posted 2017-02-08 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Surgery
Keywords: EEG electrodes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EEG Electrode Patch: The additional electrodes are modified EEG electrodes (used in clinical practice on the head already) placed in a silicone molding. These are placed lateral to the eye with the patient asleep. These are then wired to the same recording apparatus that is commonly used for recording.
  Interventions: Device: EEG Electrode Patch
- Standard Needles: The current solution to monitor eye movement during surgery is to place standard needles in the muscles surrounding the eye.
  Interventions: Device: Standard Needles

INTERVENTIONS:
Device: EEG Electrode Patch — The additional electrodes are modified EEG electrodes (used in clinical practice on the head already) placed in a silicone molding. These are placed lateral to the eye with the patient asleep. These are then wired to the same recording apparatus that we would commonly use for recording.
  Groups: EEG Electrode Patch
Device: Standard Needles — Needles are placed in the muscles surrounding the eye to measure eye movements.
  Groups: Standard Needles

SUMMARY:
For procedures involving proximity to the nerves responsible for eye movement, the need to monitor eye movement exists. The current solution is to place needles in the muscles surrounding the eye. The Investigators have invented a non-invasive electrode and software designed to monitor eye movements non-invasively. The electrode is placed on the skin on the corner of the eye and using the natural dipole of the eye, detects the horizontal and vertical movements of the eye. The Investigators would like to prove efficacy compared to the standard monitoring.

ELIGIBILITY:
Inclusion Criteria:

- Subject will be undergoing surgery involved of the nerves controlling the eye

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical patients determined by the PI
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Number of subjects with greater than 95% concordance in signal between the standard needles and EEG electrode patch | approximately 30 minutes
  The current method of measuring eye movement is to place needles in the muscles surrounding the eye. For the non-invasive method, the electrode is placed on the skin on the corner of the eye and using the natural dipole of the eye, detects horizontal and vertical movements of the eye. The signal comparison for the two methods would be a biphasic dipole representing eye movements compared to the compound muscle action potential of the invasive method.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie J Van Gompel, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials